CLINICAL TRIAL: NCT05205928
Title: Weekly Subcutaneous Semaglutide as Adjunct to Closed-loop Therapy in Type 1 Diabetes Care: a Double-blind, Cross-over, Randomized Controlled Trial
Brief Title: Weekly Subcutaneous Semaglutide as Adjunct to Closed-loop Therapy in Type 1 Diabetes Care
Acronym: SEMA-AP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Michael Tsoukas, Assistant Professor, Endocrinology & Metabolism, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022-8097
Record Dates: First submitted 2021-12-13; First posted 2022-01-25 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Type 1 Diabetes; Diabetes Mellitus, Type 1
Keywords: Insulin; Closed-loop system; GLP-1 receptor agonist; Semaglutide; Artificial Pancreas; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Insulin Resistance | interventions — Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo + closed-loop insulin system (Active Comparator)
  Interventions: Drug: Outpatient therapy: 11 weeks of drug therapy with usual treatment + 4 weeks of closed-loop therapy
- Semaglutide, Ozempic® (at maximum tolerated dose) + closed-loop insulin system (Experimental): Semaglutide is a Glucagon-Like Peptide 1 Receptor Agonist. It stimulates GLP1 in the body, which allows for increased satiety, reduced glucagon levels, delayed gastric emptying, and in some, increased insulin secretion. It is a once per week subcutaneous injection.
  Interventions: Drug: Outpatient therapy: 11 weeks of drug therapy with usual treatment + 4 weeks of closed-loop therapy

INTERVENTIONS:
Drug: Outpatient therapy: 11 weeks of drug therapy with usual treatment + 4 weeks of closed-loop therapy — The blinded drug will be used with participant's routine therapy (+ continuous glucose monitoring if not already in use) for 11 weeks with follow-up from qualified research personnel concerning pump settings, side effects, and incremental dose increase. While continuing to use the medication, there are 4 weeks of closed-loop pump therapy and drug use; glycemic outcomes will be taken from the last 4 weeks. This will be followed by laboratory and anthropometric testing, followed by 2 weeks of wash-out.

SUMMARY:
A closed-loop insulin system, also referred to as the "artificial pancreas" (AP), is made up of an insulin pump, a continuous glucose monitor, and an application communicating between the two to adjust insulin administration based on glucose control. This is meant for the treatment of type 1 diabetes. The McGill Artificial Pancreas (MAP) has been used previously in type 1 diabetes with significant benefits. Though prior studies have shown significant benefit with this system, some challenges still exist.

Semaglutide is used in type 2 diabetes and obesity; it is a once-weekly injectable medication that increases levels of a gut hormone called Glucagon-Like Peptide-1, which modifies gastric emptying, suppresses glucagon, and suppresses appetite. Though its use is not approved in type 1 diabetes in North America, it (along with similar drugs) has been used in studies as adjunctive therapy with insulin with benefits on blood sugar control. Similar medications have been used in type 1 diabetes (such as liraglutide and exenatide), but are not as strong in glucose effect even in type 2 diabetes as compared with semaglutide.

The purpose of our study is to see if semaglutide administered weekly at the maximum tolerated dose in those with type 1 diabetes will have improved glucose control (as per time in target range from continuous glucose monitoring data) compared to placebo, while using a closed-loop insulin system.

ELIGIBILITY:
Inclusion Criteria:

* A clinical diagnosis of T1D for at least one year, as per their treating diabetes physician in agreement with the primary investigator's clinical judgment (confirmatory C-peptide and antibodies will not be required)
* Glycated hemoglobin (HbA1c) up to 11% (inclusive), performed within the last 6 months prior to study inclusion
* Insulin pump use (of any modality) for minimum 3 months
* Agreement to the use of highly effective method of birth control in persons of child-bearing age (if sexually active) and active avoidance of pregnancy during the trial. Child-bearing potential refers to participants of the female sex post-menarche and have not reached menopause or have a disclosed medical condition causing sterility (e.g. hysterectomy). Post-menopausal state refers to the absence of menses for 12 months without any alternative cause.

Exclusion Criteria:

1. Current or < 2 week use of another GLP1-receptor agonist
2. Less than 2 weeks use of any anti-hyperglycemic agent other than insulin
3. Planned or ongoing pregnancy
4. Breastfeeding individuals
5. Severe hypoglycemic episode within the last 3 months, defined as an event where glucose was < 4 mmol/L resulting in seizure, loss of consciousness, or need to present to the emergency department
6. Severe diabetic ketoacidosis (DKA) within the last 6 months ("severe" referring to need to present to medical attention and requirement of intravenous insulin)
7. Prior history of acute pancreatitis, chronic pancreatitis, or gallbladder disease
8. Personal or family history of medullary thyroid cancer or multiple endocrine neoplasia type 2
9. Severe impairment of renal function with eGFR <15 mL/min/1.73 m2 (using CKD-EPI formula), measured within the last 12 months
10. Clinically significant diabetic retinopathy or gastroparesis, as per the clinical judgment of the investigator
11. History of bariatric surgery within 6 months of screening
12. Any serious medical or psychiatric illness likely to interfere with study participation as per the judgment of the investigator (e.g. cirrhosis, active cancer, decompensated schizophrenia)
13. Prior adverse reaction to GLP1-RAs
14. Body mass index ≤ 21 kg/m2
15. Regular use of hydroxyurea during the expected time of Dexcom G6 use, as this medication is known to cause inaccurate measurements (43)
16. Failure to comply to the study protocol and/or research group's recommendations (e.g. change in pump parameters, ketone measurement)
17. Inability or unwillingness to comply to safe diabetes management in the view of the study group (e.g. inappropriate treatment of hypoglycemia or lack thereof)
18. Any demonstrate of difficulty in using the iMAP system following training, as per investigator's judgment
19. Concern for safety of the participant, as per the clinical judgment of the primary investigator

**Note that for reasons of medicolegal protection for medical supervision, participants must be Canadian residents.**

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Percentage of time of plasma glucose levels spent in target range (semaglutide vs placebo) | 4 weeks
  Target range is defined to be between 3.9 and 10.0 mmol/L of placebo on closed-loop system vs semaglutide (at maximal tolerated dose) on closed-loop insulin system.

SECONDARY OUTCOMES:
Percentage of time spent in the following ranges of glucose levels between 3.9 and 7.8 mmol/L | 4 weeks
  % as per CGM data
Percentage of time spent in the following ranges of glucose levels: below 3.9 and 3.0 mmol/L | 4 weeks
  % as per CGM data
Percentage of time spent in the following ranges of glucose levels: above 7.8, 10, and 13.9 mmol/L | 4 weeks
  % as per CGM data
Mean glucose level | 4 weeks
  Defined as per CGM data, in mmol/L
Standard deviation of glucose levels as a measure of glucose variability | 4 weeks
  Defined as per CGM data, in mmol/L
Percentage coefficient of variation of glucose levels | 4 weeks
  % as per CGM data
Proportion of participants with TIR between 3.9 - 10.0 mol/L ≥ 70% | 4 weeks
  As per CGM data
Glycated hemoglobin | 15 weeks
  Blood test to assess control within last 3-4 months
Average scores between interventions based on quality of life questionnaires | 15 weeks
  These include: Type 1 Diabetes Distress Scale, Hypoglycemic Fear Survey - II, INSPIRE questionnaire for adults, Diabetes Bowel Syndrome Questionnaire, Diabetes Treatment Satisfaction Questionnaire
Blood pressure and heart rate | 15 weeks
  Body measurements as described (mmHg and beats per minutes)
Measured of body mass: weight, body mass index, waist circumference, hip circumference, waist-to-hip ratio | 15 weeks
  Measurements done at visit - weight in kilograms, body mass index as per kg/m^2, circumferences in cm
Lipid profile, specifically: LDL-cholesterol, HDL-cholesterol, triglycerides | 15 weeks
  Blood tests, in mmol/L
Biochemical analyses (exploratory) | 15 weeks
  CRP, ferritin, IL-6, Brain natriuretic peptide, TXNIP
Urine albumin-creatinine ratio | 15 weeks
  Urine test
Glucagon, C-peptide, Paracetamol absorption after mixed meal tolerance test (in first 15 participants) | 15 weeks
  Test done where beverage given and subsequent blood tests done after.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Institute of the McGill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Protocol will be included upon finalization onto the website, as well as upon request.
Supporting Information: Study Protocol

REFERENCES:
- [Derived] Pasqua MR, Doumat J, Tsoukas MA, Haidar A. Semaglutide Use With Automated Insulin Delivery in Adults With Type 1 Diabetes: Qualitative Analyses and Patient-reported Outcomes From a Randomized Controlled Trial. Can J Diabetes. 2025 Oct 30:S1499-2671(25)00367-3. doi: 10.1016/j.jcjd.2025.10.175. Online ahead of print. PMID 41175929
- [Derived] Pasqua MR, Tsoukas MA, Kobayati A, Aboznadah W, Jafar A, Haidar A. Subcutaneous weekly semaglutide with automated insulin delivery in type 1 diabetes: a double-blind, randomized, crossover trial. Nat Med. 2025 Apr;31(4):1239-1245. doi: 10.1038/s41591-024-03463-z. Epub 2025 Jan 10. PMID 39794615

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/28/NCT05205928/Prot_SAP_000.pdf